CLINICAL TRIAL: NCT04132830
Title: HIV Exposure in Utero and Metabolic Disease Risk in HIV-Negative Young Adults
Acronym: HIV HEREDITY
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lindsay Fourman, MD, Instructor in Medicine, Massachusetts General Hospital
Other Study IDs: 2019P000629
Record Dates: First submitted 2019-10-07; First posted 2019-10-21 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: HIV-exposed Uninfected
Keywords: HIV-exposed Uninfected; In Utero Exposure; Metabolic; Immune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV-Exposed Uninfected Dyads: Mothers who had HIV during pregnancy and their HIV-negative young adult offspring
  Interventions: Other: In Utero HIV Exposure
- HIV-Unexposed Uninfected Dyads: Mothers and young adults without HIV
  Interventions: Other: No In Utero HIV Exposure

INTERVENTIONS:
Other: In Utero HIV Exposure — Born to mother who had HIV infection during pregnancy.
  Groups: HIV-Exposed Uninfected Dyads
Other: No In Utero HIV Exposure — Born to mother who did not have HIV infection during pregnancy.
  Groups: HIV-Unexposed Uninfected Dyads

SUMMARY:
Globally, over 1 million babies are born to mothers with HIV each year. With the advent of prenatal antiretroviral therapy, up to 98% of these individuals may be HIV-exposed uninfected (HEU). A growing literature suggests that in utero HIV exposure - even in the absence of subsequent infection - may be associated with adverse health outcomes in infancy and childhood. However, there is little information about the long-term health implications of in utero HIV exposure later in life, such as into adulthood. In this study, for the first time, we seek to prospectively evaluate metabolic and immune indices among HEU young adults as compared to well-matched HIV-unexposed uninfected controls. This study serves as a necessary first step toward optimizing clinical care for this expanding and aging HEU population, including the implementation of novel screening and prevention strategies.

ELIGIBILITY:
INCLUSION CRITERIA:

HIV-Exposed Uninfected (HEU) Mother-Young Adult Dyads

1. Male or female young adult, 18-35 years old
2. Documentation of HIV infection in mother with date of diagnosis preceding young adult birth date
3. Negative HIV test in young adult

Control Mother-Young Adult Dyads

1. Matching to HEU dyad
2. Negative HIV test in mother and young adult

EXCLUSION CRITERIA:

All Young Adults

1. Pregnancy within 6 months or active nursing
2. Change in blood glucose or blood pressure medication within 3 months
3. Change in estrogen or testosterone therapy within 3 months
4. Chronic glucocorticoids (except steroid inhalers or creams) within 3 months
5. Antiretroviral therapy use within 6 months (i.e., prophylaxis)
6. Significant chronic illness judged by the investigator to represent a contraindication to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting mothers who had HIV during pregnancy and their HIV-negative young adult offspring (18-35 years old). We are also recruiting mothers and their young adult offspring without HIV to serve as controls.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | Baseline
Activated CD8+ T cells | Baseline
  Flow cytometry

SECONDARY OUTCOMES:
Abdominal fat mass | Baseline
  Dual-energy x-ray absorptiometry
Glucose tolerance | Baseline
  Oral glucose tolerance test
Lipids | Baseline
  Standard lipid panel (including HDL, triglycerides)
Blood pressure | Baseline
  Systolic and diastolic
Hepatic fat content | Baseline
  Transient elastography
Hepatic fibrosis | Baseline
  Transient elastography
Immune cell subsets | Baseline
  Flow cytometry
Inflammatory markers | Baseline
  ELISA
Frequency of Asthma | Baseline, Ever
DNA methylation patterns | Baseline
  Epigenome-wide analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay T Fourman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States